CLINICAL TRIAL: NCT04803110
Title: Soft Tissue Volume Changes After Immediate Implants With Two Different Techniques: Randomized Comparative Study.
Brief Title: Soft Tissue Volume Changes After Immediate Implants With Two Different Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POSTEXO
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dental Implant; Tooth Extraction; Bone Resorption
Keywords: Postextraction implant; Implant type 1; Socket-Shield; Soft Tissue volume; RCT
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: 10 receiving immediate implant placement with Socket-Shield Technique and 10 receiving immediate implant placement with complete extraction of the tooth. (n=20)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Implant with SST (SST) (Experimental): Patients who will receive immediate implant placement using the Socket-Shield Technique.
  Interventions: Procedure: Dental implant placement after tooth extraction
- Immediate Implant with biomaterial (GAP) (Active Comparator): Patients who will receive immediate implant placement using bone biomaterials to fill the gap after complete extraction of the tooth.
  Interventions: Procedure: Dental implant placement after tooth extraction

INTERVENTIONS:
Procedure: Dental implant placement after tooth extraction — Immediate implant placement after partial or complete tooth extraction.
  Other Names: Implant surgery

SUMMARY:
The aim is to comparatively evaluate the soft tissue volume changes that occur after tooth extraction and immediate dental implant placement using two different surgical techniques.

These techniques are: the Socket-Shield technique and conventional immediate placement.

The null hypothesis is that the Socket-Shield technique better maintains soft tissue volume after partial tooth extraction and immediate implant placement compared to the conventional technique.

From a sample of 20 patients, they will be divided into groups of 10 and will be randomized using the random.org program.

The soft tissue volume will be digitally recorded by intraoral scanning before tooth extraction and 6 months later.

The soft tissue dimensional changes produced will be digitally evaluated and statistically analyzed.

DETAILED DESCRIPTION:
After tooth extraction, the supporting tissues, bone and mucosa will undergo a loss of volume associated with the loss of the cementum-periodontal ligament-bone attachment complex.

This alteration in volume can affect aesthetic results, especially when the tooth involves the anterior area, where the alveolar bone is narrower.

To compensate for the lost volume loss, some authors promote delayed implant placement, which would facilitate soft tissue management after healing.

The conventional immediate implant placement technique proposes the use of bone regeneration biomaterials in the space between the implant wall and the residual vestibular bone. The aim of this technique is to compensate for this bone resorption, thus improving the aesthetic results. In the same sense of compensating for the resorption that will occur, some authors recommend the use of soft tissue grafts in the same operative act of extraction and placement of the immediate implant.

Some years ago, some authors presented the technique of partial extraction of the tooth as an alternative to the conventional technique of immediate implant placement after extraction with the aim of avoiding or minimising this resorption. The technique consists of leaving a piece of tooth (shield) inserted in the vestibular alveolar bone area so that the resorption process is slowed down.

The presence of bone between the dentine wall of the tooth fragment and the implant has been demonstrated in both animal and ex-vivo histological studies.

From a clinical point of view, the Socket-Shield or partial extraction technique has been shown to maintain the vestibular volume in post-extraction implants placed using this technique in both posterior and anterior areas with high aesthetic compromise, maintaining adequate clinical values and patient satisfaction.

On the other hand, a 2015 systematic review, comparing immediate and delayed implantation techniques, reports no significant differences between the two, especially at the soft tissue level, although it mentions a lack of quality in the RCTs analysed.

A 2017 randomized clinical trial compared the conventional immediate implant placement technique with the delayed or early implantation technique, advising against the former when aesthetics were compromised and limiting it to well-selected cases.

In contrast, another more recent randomized clinical trial found no aesthetic, clinical or radiographic differences between the two techniques, and reported similar levels of patient satisfaction.

Likewise, a higher rate of early failure has been found in the immediate implantation technique, mentioning the lack of randomised clinical studies comparing both techniques, especially in terms of soft tissue volume changes.

A recent randomised clinical study comparing the Socket-Shield technique with the conventional implant placement technique found better levels of marginal bone and pink aesthetic assessment in the former, considering it a safe and feasible technique in the anterior sector.

Given the lack of evidence in the literature, there is a palpable need for clinical studies to compare the best technique and/or timing of implant placement after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring single tooth extraction in lateral or anterior areas of the upper jaw.
* Teeth that do not present alteration or loss of the vestibular bone table.

Exclusion Criteria:

* Patients in whom surgical intervention is contraindicated.
* Teeth with alteration or loss of the vestibular bone table.
* Teeth with marginal recession >2mm.
* Early or delayed failure of the implant placed with any of the three techniques.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue volume | 6 months
  Soft tissue volume changes after tooth extraction

SECONDARY OUTCOMES:
Surgery pain perception by Numerical Rating Scale | Just after surgery
  Pain perception by the patient during surgical procedure, being 0 no pain at all, 1-3 mild discomfort, 4-7 moderate pain and 7-10 intense pain.
Surgery satisfaction of the patient by Numerical Rating Scale | Just after surgery
  Patients satisfaction after surgery, being 0 not satisfied at all, and 10 very satisfied
General satisfaction of the patient by Numerical Rating Scale | 6 months after the beginning of treatment
  Patients general satisfaction 6 months after the beginning of treatment, being 0 not satisfied at all, and 10 very satisfied
Esthetic satisfaction of the patient by Numerical Rating Scale | 3 months after after crown placement
  Patients esthetic satisfaction 3 months after crown placement, being 0 not satisfied at all, and 10 very satisfied
Function satisfaction of the patient by Numerical Rating Scale | 3 months after after crown placement
  Patients function satisfaction 3 months after crown placement, being 0 not satisfied at all, and 10 very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, Principal Investigator — Aula Dental Avanzada
Locations (1):
- Clínica Dental Esteve, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
No plan to share with other researches.

REFERENCES:
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Chen ST, Buser D. Esthetic outcomes following immediate and early implant placement in the anterior maxilla--a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:186-215. doi: 10.11607/jomi.2014suppl.g3.3. PMID 24660198
- [Background] Lee CT, Chiu TS, Chuang SK, Tarnow D, Stoupel J. Alterations of the bone dimension following immediate implant placement into extraction socket: systematic review and meta-analysis. J Clin Periodontol. 2014 Sep;41(9):914-26. doi: 10.1111/jcpe.12276. Epub 2014 Jul 23. PMID 24894299
- [Background] Buser D, Chen ST, Weber HP, Belser UC. Early implant placement following single-tooth extraction in the esthetic zone: biologic rationale and surgical procedures. Int J Periodontics Restorative Dent. 2008 Oct;28(5):441-51. PMID 18990995
- [Background] Seyssens L, De Lat L, Cosyn J. Immediate implant placement with or without connective tissue graft: A systematic review and meta-analysis. J Clin Periodontol. 2021 Feb;48(2):284-301. doi: 10.1111/jcpe.13397. Epub 2020 Nov 20. PMID 33125754
- [Background] Hurzeler MB, Zuhr O, Schupbach P, Rebele SF, Emmanouilidis N, Fickl S. The socket-shield technique: a proof-of-principle report. J Clin Periodontol. 2010 Sep;37(9):855-62. doi: 10.1111/j.1600-051X.2010.01595.x. PMID 20712701
- [Background] Mitsias ME, Siormpas KD, Kotsakis GA, Ganz SD, Mangano C, Iezzi G. The Root Membrane Technique: Human Histologic Evidence after Five Years of Function. Biomed Res Int. 2017;2017:7269467. doi: 10.1155/2017/7269467. Epub 2017 Nov 22. PMID 29333449
- [Background] Baumer D, Zuhr O, Rebele S, Schneider D, Schupbach P, Hurzeler M. The socket-shield technique: first histological, clinical, and volumetrical observations after separation of the buccal tooth segment - a pilot study. Clin Implant Dent Relat Res. 2015 Feb;17(1):71-82. doi: 10.1111/cid.12076. Epub 2013 Apr 30. PMID 23631704
- [Background] Baumer D, Zuhr O, Rebele S, Hurzeler M. Socket Shield Technique for immediate implant placement - clinical, radiographic and volumetric data after 5 years. Clin Oral Implants Res. 2017 Nov;28(11):1450-1458. doi: 10.1111/clr.13012. Epub 2017 Mar 23. PMID 28333394
- [Background] Barbisan A, Dias CS, Bavia PF, Sapata VM, Cesar-Neto JB, Silva CO. Soft Tissues Changes After Immediate and Delayed Single Implant Placement in Esthetic Area: A Systematic Review. J Oral Implantol. 2015 Oct;41(5):612-9. doi: 10.1563/AAID-JOI-D-13-00095. Epub 2014 Jan 29. PMID 24475930
- [Background] Tonetti MS, Cortellini P, Graziani F, Cairo F, Lang NP, Abundo R, Conforti GP, Marquardt S, Rasperini G, Silvestri M, Wallkamm B, Wetzel A. Immediate versus delayed implant placement after anterior single tooth extraction: the timing randomized controlled clinical trial. J Clin Periodontol. 2017 Feb;44(2):215-224. doi: 10.1111/jcpe.12666. Epub 2017 Jan 31. PMID 27978602
- [Background] Huynh-Ba G, Hoders AB, Meister DJ, Prihoda TJ, Mills MP, Mealey BL, Cochran DL. Esthetic, clinical, and radiographic outcomes of two surgical approaches for single implant in the esthetic area: 1-year results of a randomized controlled trial with parallel design. Clin Oral Implants Res. 2019 Aug;30(8):745-759. doi: 10.1111/clr.13458. Epub 2019 Jun 7. PMID 31099929
- [Background] Cosyn J, De Lat L, Seyssens L, Doornewaard R, Deschepper E, Vervaeke S. The effectiveness of immediate implant placement for single tooth replacement compared to delayed implant placement: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:224-241. doi: 10.1111/jcpe.13054. PMID 30624808
- [Background] Bramanti E, Norcia A, Cicciu M, Matacena G, Cervino G, Troiano G, Zhurakivska K, Laino L. Postextraction Dental Implant in the Aesthetic Zone, Socket Shield Technique Versus Conventional Protocol. J Craniofac Surg. 2018 Jun;29(4):1037-1041. doi: 10.1097/SCS.0000000000004419. PMID 29489581